CLINICAL TRIAL: NCT00912262
Title: A Randomized, Single Blind Study to Investigate the Tolerability and Effects on Epidermal Nerve Fiber Density of Multiple Low-Concentrations of Capsaicin Topical Liquid NGX-1998 in Healthy Volunteers
Brief Title: A Study to Investigate the Tolerability and Effects on Epidermal Nerve Fiber Density of Multiple Low-Concentrations of NGX-1998 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C203
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Pain
Keywords: Analgesics; Capsaicin
MeSH Terms: conditions — Pain

ARMS (1):
- Low and High Concentration Capsaicin Topical Liquids (Active Comparator)
  Interventions: Drug: Capsaicin Topical Liquid

INTERVENTIONS:
Drug: Capsaicin Topical Liquid

SUMMARY:
The purpose of this single-blinded study in healthy volunteers is to select a Low-Concentration Capsaicin Topical Liquid (LC-CTL) to serve as a control formulation in the further clinical development of Capsaicin Topical Liquid, NGX-1998 (10% w/w). The goal is to identify a low concentration formulation that will not reduce ENFD in healthy normal volunteers when compared to NGX-1998 (10% w/w) but would still produce some local capsaicin-related application site responses (e.g. erythema, heat sensation or pain) when applied.

DETAILED DESCRIPTION:
This is a randomized, single center, single-blind controlled study in up to 36 healthy volunteers. Each subject will be dosed at four application sites, 7 by 7 cm in size, located n the distal and proximal anterior medial thigh areas. At two sites, subjects will receive 15-minute treatments of a LC-CTL (1%, 0.3%, 0.1%, 0.003% or 0.001% w/w). At the remaining two sites, subjects will receive 15-minute treatments of NGX-1998 (10% w/w) and a control liquid (CTL-V (0%)). The volume applied at each application site is estimated to be 7 mcl per cm2 and hence the total volume of approximately 300 mcl of LC-CTL (all concentrations), NGX-1998 (10% w/w) and CTL-V (0%) applied at each site application will be sufficient to evenly wet the surface.

The top or bottom section of each application site will be pre-treated with lidocaine 2.5% / prilocaine 2.5% topical anesthetic cream. These sections are also the sections where the skin punch biopsies will be taken. The biopsy will be obtained from these sections as it is anticipated that subsequent clinical trials in patients will use pre-treatment with a topical anesthetic. However, only the toop or bottom sections will be pre-treated with this topical anesthetic so that pre-treatment with the topical anesthetic cream does not interfere with tolerability assessments.

The pharmacodynamic effects of nerve fiber density and function will be evaluated by immunohistochemical staining of biopsied tissue from the treatment area. Skin punch biopsies at all four application sites will be obtained to evaluate ENFD at 7 days post-application.

Safety and tolerability will be evaluated by continuous monitoring of adverse events (AEs0 and periodic assessments of clinical laboratory parameters, vital signs, physical examinations, dermal assessments, and pain associated with treatment.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, subjects must meet all of the Inclusion Criteria:

* 18 to 40 years of age, inclusive. Male and female subjects.
* Be in good health
* Have intact, unscarred skin over the thighs
* Agree not to use topically-applied products containing non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics, steroids or capsaicin anywhere on the thighs for the duration of the study
* Female subjects of child bearing potential must not be breast-feeding and must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test performed within 7 days prior to the Application Visit (Day 0)
* All subjects, including early terminations, must be willing to use effective methods of birth control and/or refrain from participating in a conception process during the study and for 30 days following experimental drug exposure
* Subjects must be willing and able to comply with protocol requirements for the duration of study participation. Requirements include but are not limited to attending all study visits and refraining from extensive travel during study participation
* Subjects must sign an informed consent form that has been approved by the Investigator's Institutional Review Board (IRB) to participate in this study

Exclusion Criteria:

* Any dermatological condition(s) that in the judgment of the Principal Investigator has the potential to disrupt skin integrity, healing, or alter sensory function on the thighs.
* Any skin infection, skin irritation (e.g., poison oak), history of eczema, trauma or burn (including sunburn) on the thighs within 30 days preceding the Application Visit (Day 0).
* Any medical history of painful conditions, surgery, or injury involving or affecting the thighs, including but not limited to prior orthopedic surgery, lumbosacral disc disease, sciatica, and hip or femur fracture.
* Any medical history of known or suspected body system abnormalities, including but not limited to diabetes, hypothyroidism, asthma or any form of peripheral or central nervous system disease.
* Subjects with congenital, idiopathic, or drug-induced methemoglobinemia.
* Use of any systemic medications that interact with the peripheral nervous system, including beta adrenergic blockers, alpha adrenergic blockers, anticonvulsant drugs, antidepressant drugs or opioids within 30 days prior to the Application Visit (Day 0).
* Current use of any class III anti-arrhythmic drugs (eg, amiodarone, bretylium, sotalol, dofetilide).
* Use of any topically-applied product, including prescription or over the-counter (OTC) analgesic creams/lotions/patches, non steroidal anti-inflammatory drugs, counterirritants, local anesthetics, steroids or capsaicin on the thighs within 30 days preceding the Application Visit (Day 0).
* Currently taking any prescription medication except for oral, transdermal or injected contraceptives.
* Requirement for ongoing or periodic pain medication for any chronic or recurrent medical condition. Refer to Section 3.4 for additional information about concomitant medications.
* Participation in another drug research study within 30 days preceding the Application Visit (Day 0).
* Diagnosis of human immunodeficiency virus (HIV) infection, according to medical history and/or self-report; or Positive test result on the HIV-1 blood test performed at the Screening Visit (ICMA with Western Blot confirmation).
* History or current substance abuse including alcoholism/alcohol abuse.
* Positive test result on the urine drug screen for barbiturates, benzodiazepines, tricyclic anti-depressants, propoxyphene, opioids, cannabis, phencyclidine (PCP), cocaine and amphetamines performed at the Screening Visit.
* History of hypersensitivity to capsaicin (i.e., chili peppers or OTC capsaicin products), local anesthetics (including lidocaine and prilocaine) or any components of the Capsaicin Topical Liquids, Cleansing Gel or the lidocaine 2.5% / prilocaine 2.5% topical anesthetic cream.
* Any clinically-significant abnormal laboratory test at the Screening Visit.
* Clinically-significant abnormal 12-Lead ECG at the Screening Visit

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-06; Study Completion 2008-11

PRIMARY OUTCOMES:
To assess the potential differences in the effects of 15-minute treatments of several Low-Concentration Capsaicin Topical Liquids, compared to 15-minute treatments of NGX-1998 and a control, Capsaicin Topical Liquid Vehicle, as quantified by Protein Gene

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Tobias, MD, Study Director — NeurogesX
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States